CLINICAL TRIAL: NCT02589379
Title: The Value of Endoscopic Ultrasound Elastography for Prediction of Pancreatic Fistula in Patients Undergoing Pancreatic Resection for Benign or Malignant Disease
Brief Title: Ultrasound Elastography for Prediction of Postoperative Pancreatic Fistula
Acronym: PMPPOPF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Mickael Lesurtel, Professor, MD, PhD, University of Zurich
Other Study IDs: POPF-0134
Record Dates: First submitted 2015-10-09; First posted 2015-10-28 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Pancreatic Fistula
Keywords: postoperative pancreatic fistula; soft and hard pancreas
MeSH Terms: conditions — Pancreatic Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Non-tumorous pancreatic tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pancreatic Resection: All consecutive patients undergoing pancreatic resection for benign or malignant disease and meet inclusion criteria.
  Interventions: Procedure: Pancreatic Resection

INTERVENTIONS:
Procedure: Pancreatic Resection — Endoscopic ultrasound elastography, intraoperative ultrasound elastography and magnet resonance imaging to asses pancreatic stiffness prior to pancreatic resection

SUMMARY:
The purpose of this study is to assess the value of preoperative objective modalities such as endoscopic ultrasound elastography and magnet resonance imaging in predicting development of postoperative pancreatic fistula in patients undergoing pancreatic surgery for benign or malignant disease.

DETAILED DESCRIPTION:
One of the most generally accepted causes of postoperative pancreatic fistula (POPF) is soft texture of the pancreas. The stiffness of organs depends on histologic features such as content of fat, fibrotic tissue and micro vascular structures. Yet, pancreatic stiffness was evaluated only subjectively. Endoscopic ultrasonography (EUS) and magnetic resonance imaging (MRI) may allow objective quantification of pancreatic stiffness prior to surgery.

Endoscopic ultrasound elastography (EUE) is based on real-time Doppler technology. Image colors are derived from vibration patterns which depend on the stiffness of a specific region of the investigated organ. The retrieved images could be converted into numeric matrix using a specially designed program.

Magnetic resonance imaging (MRI) is a non-invasive method for quantitatively assessing the mechanical properties of tissues based on fat tissue content.

In this trial the investigators will assess at first the value of EUE and MRI in predicting development of postoperative pancreatic fistula and in a next step the value EUE and MRI as an objective method in prediction of pancreatic stiffness.

ELIGIBILITY:
Inclusion Criteria:

* Adult (more than 18 years) with resectable pancreatic lesion(s)

Exclusion Criteria:

* Total pancreatectomy
* Unresectable pancreatic lesion(s)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing pancreatic resection for benign or malignant disease
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2015-07; Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
POPF rate (in %) as defined by the International Study Group on Pancreatic Fistula (ISGPF) in the soft versus hard pancreas group based on the median EUE stiffness measurements generated by values derived from hue histograms. | within the 30 days after surgery

SECONDARY OUTCOMES:
Pearson correlation coefficient between preoperative EUE measurements of pancreatic stiffness generated by values derived from hue histograms with the fat content (in %) of the resected specimen on histology. | within the 30 days after surgery
Pearson correlation coefficient between preoperative EUE measurements of pancreatic stiffness generated by values derived from hue histograms with intra-operative ultrasound elastography measurements generated by values derived from hue histograms. | within the 30 days after surgery
Postoperative pancreatic fistula rate (in %) as defined by the ISGPF in the soft versus hard pancreas group based on the median MRI fat measurement (in %) on histology. | within the 30 days after surgery
Pearson correlation coefficient between preoperative MRI measurements of pancreatic fat (in %) with the fat content (in %) of the resected specimen on histology. | within the 30 days after surgery
Postoperative pancreatic fistula rate (in %) as defined by the ISGPF in the soft versus hard pancreas group based on the surgeons assessment of stiffness on a visual analogue scale from soft (0) to hard (10) intraoperatively. | within the 30 days after surgery
Pearson correlation coefficient between the two surgeons assessing pancreatic stiffness intraoperatively. | within the 30 days after surgery
Intraclass correlation coefficient of the all measurements derived from EUE, IUE, MRI, surgeons assessment and histology. | within the 30 days after surgery
  within the 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Petrowsky, Prof, MD, Study Chair — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Result] Bassi C, Dervenis C, Butturini G, Fingerhut A, Yeo C, Izbicki J, Neoptolemos J, Sarr M, Traverso W, Buchler M; International Study Group on Pancreatic Fistula Definition. Postoperative pancreatic fistula: an international study group (ISGPF) definition. Surgery. 2005 Jul;138(1):8-13. doi: 10.1016/j.surg.2005.05.001. PMID 16003309
- [Result] Lin JW, Cameron JL, Yeo CJ, Riall TS, Lillemoe KD. Risk factors and outcomes in postpancreaticoduodenectomy pancreaticocutaneous fistula. J Gastrointest Surg. 2004 Dec;8(8):951-9. doi: 10.1016/j.gassur.2004.09.044. PMID 15585382
- [Result] Mathur A, Pitt HA, Marine M, Saxena R, Schmidt CM, Howard TJ, Nakeeb A, Zyromski NJ, Lillemoe KD. Fatty pancreas: a factor in postoperative pancreatic fistula. Ann Surg. 2007 Dec;246(6):1058-64. doi: 10.1097/SLA.0b013e31814a6906. PMID 18043111
- [Result] Nathan H, Cameron JL, Goodwin CR, Seth AK, Edil BH, Wolfgang CL, Pawlik TM, Schulick RD, Choti MA. Risk factors for pancreatic leak after distal pancreatectomy. Ann Surg. 2009 Aug;250(2):277-81. doi: 10.1097/SLA.0b013e3181ae34be. PMID 19638926
- [Result] Saftoiu A, Vilmann P, Gorunescu F, Janssen J, Hocke M, Larsen M, Iglesias-Garcia J, Arcidiacono P, Will U, Giovannini M, Dietrich CF, Havre R, Gheorghe C, McKay C, Gheonea DI, Ciurea T; European EUS Elastography Multicentric Study Group. Efficacy of an artificial neural network-based approach to endoscopic ultrasound elastography in diagnosis of focal pancreatic masses. Clin Gastroenterol Hepatol. 2012 Jan;10(1):84-90.e1. doi: 10.1016/j.cgh.2011.09.014. Epub 2011 Oct 1. PMID 21963957
- [Result] Sato N, Yamaguchi K, Chijiiwa K, Tanaka M. Risk analysis of pancreatic fistula after pancreatic head resection. Arch Surg. 1998 Oct;133(10):1094-8. doi: 10.1001/archsurg.133.10.1094. PMID 9790207
- [Result] Schafer M, Mullhaupt B, Clavien PA. Evidence-based pancreatic head resection for pancreatic cancer and chronic pancreatitis. Ann Surg. 2002 Aug;236(2):137-48. doi: 10.1097/00000658-200208000-00001. PMID 12170018
- [Result] Watanabe H, Kanematsu M, Tanaka K, Osada S, Tomita H, Hara A, Goshima S, Kondo H, Kawada H, Noda Y, Tanahashi Y, Kawai N, Yoshida K, Moriyama N. Fibrosis and postoperative fistula of the pancreas: correlation with MR imaging findings--preliminary results. Radiology. 2014 Mar;270(3):791-9. doi: 10.1148/radiol.13131194. Epub 2013 Nov 8. PMID 24475834
- [Result] Yeh TS, Jan YY, Jeng LB, Hwang TL, Wang CS, Chen SC, Chao TC, Chen MF. Pancreaticojejunal anastomotic leak after pancreaticoduodenectomy--multivariate analysis of perioperative risk factors. J Surg Res. 1997 Feb 1;67(2):119-25. doi: 10.1006/jsre.1996.4974. PMID 9073557